CLINICAL TRIAL: NCT05668507
Title: Using a Virtual Care Platform to Deliver Peer-led Mental Health Support to Rural and Remote Communities in BC: a Randomized Wait-list Controlled Trial of the REACHOUT Intervention
Brief Title: REACHOUT Mental Health Support Mobile App
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Brain Canada (Other)
Responsible Party: Principal Investigator, Tricia Tang, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H22-02196
Record Dates: First submitted 2022-12-08; First posted 2022-12-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Type1diabetes
Keywords: mental health; type 1 diabetes; peer support; technology
MeSH Terms: conditions — Psychological Well-Being; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the intervention group (access to the mobile app/support program right away) or the wait-list control group (access granted to the mobile app/support program after 6 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REACHOUT (Experimental): The REACHOUT intervention arm will receive access to the REACHOUT mobile app through which they will be able to review profiles of Peer Supporters and connect with one of their choosing. They will also have access to the other app features including a 24/7 chat room and face-to-face support via virtual happy hours. Participants will complete questionnaires (baseline, 1 month, 3 months, 6 months) and a blood draw (baseline and 6 months). Monetary compensation will be provided for their time and effort.
  Interventions: Behavioral: REACHOUT Virtual Mental Health Support
- Wait-list (No Intervention): The wait-list control group will receive access to the mobile app/support program after six (6) months. They will complete questionnaires and a blood draw at baseline and 6 months. Monetary compensation will be provided for their time and effort.

INTERVENTIONS:
Behavioral: REACHOUT Virtual Mental Health Support — REACHOUT is a mobile app which delivers peer-led mental health support to adults with type 1 diabetes. The mobile app has three support features:
  1. One-on-one support delivered by a Peer Supporter. Participants will be able to review Peer Supporter profiles and connect with one of their choosing.
  2. Group support delivered via a 24/7 chat room
  3. Face to face support delivered via virtual happy hours
  Arms: REACHOUT

SUMMARY:
The purpose of this study is to investigate the effectiveness of participation in a 6-month peer-led mental health support program, delivered via a mobile app (REACHOUT), to adults with type 1 diabetes compared to a wait-list control condition. Participants will connect with a Peer-Supporter (an adult with type 1 diabetes trained in providing mental health support), and have access to the app features including a 24/7 chat room and face-to-face support delivered via virtual happy hours.

DETAILED DESCRIPTION:
REACHOUT is a mobile app which delivers peer-led mental health support to adults with type 1 diabetes. The mobile app has three support features:

1. One-on-one support delivered by a Peer Supporter

   Peer Supporters are adults with type 1 diabetes who will be trained on providing support to other adults with type 1 diabetes on the app ("the participants"). Participants will be able to go through the peer supporter library, review their profiles, and choose their peer supporter.
2. Group support delivered via a 24/7 chat room

   Peer Supporters and participants on the app will be able to chat 24/7 in the chat room about any topic ranging from feedback on new devices to traveling with diabetes. The chat room is monitored by healthcare professionals including a registered nurse and registered psychologist.
3. Face to face support delivered via virtual happy hours

Virtual happy hours are educational presentations/discussions led by either a Peer Supporter or healthcare professional on topics related to diabetes.

Participants will be randomly assigned to the intervention group or the wait-list control group. The intervention group will be given access to the mobile app right away and the wait-list control group will be given access to the mobile app after six months.

The intervention is 6 months long. All participants and Peer Supporters will go through an assessment at the start and end of the program. The assessment includes a blood draw to measure hemoglobin A1c, and questionnaires measuring diabetes distress, perceived social support, depressive symptoms, resilience, quality of life, and costs related to diabetes. There will also be questionnaires throughout the program including at 1-month and 3-months. Participants and Peer Supporters who own a Dexcom G6 continuous glucose monitor (CGM) will be asked if they would like to share their CGM data.

ELIGIBILITY:
Inclusion Criteria:

* have type 1 diabetes (T1D)
* be 19 years or older
* reside in one of the targeted health authorities in British Columbia (Fraser Health, Island Health, Northern Health, and Interior Health Authorities)
* be English proficient
* have an average diabetes distress (DD) Subscale Score ≥ 2
* have access to the internet and/or a smartphone.

Exclusion Criteria:

* Participants with a pre-existing mental health condition, multiple co-morbidities, substance use challenges, and or any other condition that may prevent meaningful participation may not participate in this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Distress | 0, 6 month(s)
  Diabetes Distress will be measured by the Type 1 Diabetes Distress Scale (T1D-DDS). This scale contains 28 items that people with type 1 diabetes may find distressing. Participants rate each item on a scale from 1 indicating Not a Problem to 6 indicating a Very Serious Problem. There are seven subscales including powerlessness, management distress, hypoglycemia distress, negative social distress, eating distress, physician distress, and family/friends distress. Overall and subscale scores are calculated by taking the mean of items in the overall or subscale. A higher score indicates higher diabetes distress.

SECONDARY OUTCOMES:
Change in Perceived social support | 0, 6 month(s)
  Perceived Social Support will be assessed using the Diabetes-Specific Perceived Social Support Scale. This scale presents a list of ways that people give and receive support, and asks participants to indicate the degree to which each statement is true for them. Participants may rate each item from 0 indicating No Support to 4 indicating a Great Deal of Support. A higher score indicates higher perceived social support.
Change in Depressive Symptom Severity | 0, 6 month(s)
  Depressive Symptom Severity will be assessed using the Personal Health Questionnaire 8 (PHQ-8). This questionnaire asks participants how bothered they have been by various problems over the past two weeks. Participants rate each item from 0 indicating Not At All to 3 indicating Nearly Every Day. A total score is calculated by adding up the ratings for each item. A higher score indicates higher depressive symptom severity.
Change in Resilience | 0, 6 month(s)
  Resilience will be assessed by the Diabetes Strengths and Resilience (DSTAR) Measure for Emerging Adults. The scale presents a list of items that people with diabetes sometimes think. Items are scored on a 5-point Likert scale from never "1" to almost always "5". A total score is calculated by taking a sum of all items. A higher score indicates higher resilience.
Change in Diabetes-Specific Quality of Life | 0, 6 month(s)
  Diabetes-Specific Quality of Life will be measured by the Type 1 Diabetes Activities and Living (T1DAL). The survey questions ask participants what their life is like with diabetes including what is going well for them or what they could use more help with. There are different variations of the questionnaire for each of the following age cohorts: 18 - 25 years old, 26 - 45 years old, 46 - 60 years old, > 60 years old. Participants answer each item with the following options: (1) No, not at all true; (2) No, not very true; (3) Sometimes true, sometimes not true; (4) Yes, a little true; (5) Yes, very true.
Change in Health-Related Quality of Life | 0, 3, 6 month(s)
  Health-Related Quality of Life will be measured by the EuroQol-5D-5 level version (EQ-5D-5L), which asks questions regarding general health. Participants are asked to choose from a variety of statements for each question which best describes their health.
Change in Quality Adjusted Life year (QALY) | 0, 3, 6 month(s)
  Change Quality Adjusted Life Year (QALY) will be estimated using the Visual Analogue Scale (VAS) of the EuroQol-5D-5 level version (EQ-5D-5L). The VAS asks participants to self-rate their health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Change in Health Related Costs | 0, 3, 6 month(s)
  Change in Health Related Costs will be measured by the Health Resource Utilization Questionnaire (HRU). This questionnaire asks a series of questions regarding health resource utilization and costs patients may have incurred.
Change in Hemoglobin A1c | 0, 6 month(s)
  Hemoglobin A1c (HbA1c) will be measure via blood collection
Change in % Time in Range | 14 days before and after each participant's baseline and 6-month assessments, respectively
  In British Columbia, the continuous glucose monitor (CGM) brands that are covered by provincial health care are the Dexcom G6, G7, and Freestyle Libre 2. As such, we will request to collect % time in range data from all participants who are using this CGM. Because the CGMs are pre-calibrated by the factory, participants do not need to self-calibrate. CGM units will be retrieved by the research team using Dexcom Clarity software (Dexcom, San Diego, CA), LibreView. We will also request participants who are using Glooko to share their data with us by uploading their data onto their Glooko account. In order to understand blood glucose fluctuations, we will collect 14 days of CGM glucose data at two timepoints: 1) baseline and 2) 6 months. The first day will be considered as the date of the baseline and 6-month assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Tricia S Tang, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada